CLINICAL TRIAL: NCT02786017
Title: The Safety and Efficacy Assessment of Injectable Collagen Scaffold™ Combined With Human Umbilical Cord-derived Mesenchymal Stem Cells (HUC-MSCs) Transplantation in Patients With Decompensated Cirrhosis
Brief Title: Injectable Collagen Scaffold™ Combined With HUC-MSCs Transplantation for Patients With Decompensated Cirrhosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAS-XDA-DC/IGDB
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2016-04

CONDITIONS: Decompensated Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional therapy (Sham Comparator)
  Interventions: Biological: Conventional therapy
- Injectable Collagen Scaffold + HUC-MSCs (Experimental)
  Interventions: Biological: Injectable Collagen Scaffold + HUC-MSCs

INTERVENTIONS:
Biological: Conventional therapy — Patients will receive the conventional therapy.
  Arms: Conventional therapy
Biological: Injectable Collagen Scaffold + HUC-MSCs — Injectable collagen scaffold combined with HUC-MSCs was injected into left lateral segment, left medial segment, right anterior segment, right posterior segment and caudate lobe under B-mode ultrasound supervision, respectively. The total amount of HUC-MSCs was 5*10^8.
  Arms: Injectable Collagen Scaffold + HUC-MSCs

SUMMARY:
The purpose of this study is to assess the safety and efficacy of injectable collagen scaffold combined with human umbilical cord-derived mesenchymal stem cells (HUC-MSCs) transplantation in patients with Decompensated Cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

1. Subjects who are decompensated cirrhosis of any cause.
2. Subjects are repeated exacerbations despite treatment and hospitalized more than once within one year because of complications of cirrhosis, (e.g., massive ascites, spontaneous bacterial peritonitis, gastrointestinal bleeding or hepatic encephalopathy).
3. Need intermittent plasma albumin and oral diuretics supplement.
4. Serum albumin <35 g/L, total bilirubin<170 μmol/L, prothrombin activity >30% (prothrombin time <20 s), moderate or mild ascites, spontaneous bacterial peritonitis and hepatic encephalopathy have been cured, Child-pugh score ≥7.
5. Peripheral blood hemoglobin concentration> 70g/L，platelet count > 3 × 10^9/L, hematocrit (HCT) level>0.25.
6. No gastrointestinal bleeding during the last one month before enrolment.
7. Patient has no conditional to undergo orthotopic liver transplantation (OLT).
8. Willing to sign informed consent.

Exclusion Criteria:

Participants CANNOT meet any of the following criteria:

1. The presence of hepatocellular carcinoma (HCC) or other malignant tumors.
2. Complicated with gastrointestinal bleeding, spontaneous bacterial peritonitis, hepatic encephalopathy, hepatorenal syndrome and acute exacerbation of infection.
3. Presence of severe comorbid diseases (e.g., severe renal, respiratory, cardiac or blood disease).
4. Pregnant or lactating women.
5. Allergy to G-CSF, contrast agents and anticoagulants.
6. Alcoholism or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of liver function measured by change in the model for end-stage liver disease (MELD) score | 1 week, 2 week, 1, 3, 6, 12, 24 month after intervention

SECONDARY OUTCOMES:
Improvement of liver function measured by change in Child-Pugh score | 1 week, 2 week, 1, 3, 6, 12, 24 month after intervention
Change in clinical laboratory parameters of liver function | 1 day, 3 day, 1 week, 2 week, 1, 3, 6, 12, 24 month after intervention
  The liver function tests included serum Albumin (Alb), Cholesterol, Cholinesterase (CHE), prothrombin activity.
30-Day Survival | 30 days
  Patients surviving more than 30 days after study registration.
Change in the size of liver and spleen and inner diameter of spleen portal venous | 1 week, 2 week, 1, 3, 6, 12, 24 month after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D, Principal Investigator — Chinese Academy of Sciences
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China